CLINICAL TRIAL: NCT02938039
Title: I-Gel vs Ambu Laryngeal Mask Airways in Infants and Children Undergoing Surgical Procedures: A Randomized Clinical Trial
Brief Title: I-Gel vs Ambu Laryngeal Mask Airways in Infants and Children Undergoing Surgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr Abdulrahman Alzahem, Associate Professor and Consultant, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E14-1153
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Laryngeal Masks
Keywords: laryngeal airways; infants; neonates; children; anesthetized

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambu LMA (Active Comparator): Ambu Laryngeal Mask Airway device of different sizes for age
  Interventions: Device: Ambu LMA
- I-Gel LMA (Active Comparator): I-Gel Laryngeal Mask Airway device of different sizes for age
  Interventions: Device: I-Gel LMA

INTERVENTIONS:
Device: Ambu LMA — Ambu Laryngeal Mask Airways
  Arms: Ambu LMA
Device: I-Gel LMA — I-Gel Laryngeal Mask Airways
  Arms: I-Gel LMA

SUMMARY:
This study will guide the anesthetists regarding the appropriate selection of the LMA in neonatal age group based on scientific basis.

This study will add up to existing literature about the safety of LMA usage in neonates and infants. Furthermore it may shed some light on which LMA type will be more feasible and effective for neonatal/ infants usage.

DETAILED DESCRIPTION:
Laryngeal mask airways (LMAs) are in practice of anesthesia since early 1980s. Pediatric and neonatal patients (including ex-premature) have also been benefited by the use of LMA. There are many advantages of LMA over endotracheal tube (ETT) in pediatric patients like ease of insertion, securing airway rapidly, avoidance of muscle relaxants, reduced incidence of sore throat, post operative hoarseness and coughing at the time of extubation, greater hemodynamic and intraocular pressure (IOP) stability. LMA has been recognized internationally in control of airway in difficult and failed intubation.

There are different types of pediatric LMAs available e.g. I-gel, ProSeal, LMA supreme, LMA classic, LMA unique, LarySeal and Ambu. These devices differ morphologically from each other (silicone, polyvinyl chloride or soft gel). There have been several randomized controlled studies comparing different LMAs in adults, however, the literature is sparse in which such comparison has been made in patients with weight 10 kg or below.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical procedures
* No muscle relaxant agents
* No other comorbidities

Exclusion Criteria:

* Emergency surgical procedures
* Full stomach
* Subjects with upper respiratory tract infection
* Failed caudal block

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Airway Leak Pressure | 17 months
  It will be measured in mmHg unit and the expiratory valve will be closed with a fresh gas flow of 3 l.min-1 until an audible leak is heard, airway pressure will not be allowed to exceed 25 cmH2O), and then released completely

SECONDARY OUTCOMES:
Effective airway time | 18 months
  It will be measured in seconds unit , and The time for successful insertion will be measured from the moment the facemask will be removed until attainment of first capnography upstroke after insertion
Ease of insertion | 18 months
  The ease of placement of LMA will be assessed using a subjective scale of 1-4 (1 = no resistance and no maneuvers, 2 = mild resistance and one maneuver, 3 = moderate resistance and more than one maneuver, 4 = inability to place the device)
Success at first attempt | 18 months
  The insertion will be labelled as a 'failure' if the device could not be successfully placed within two attempts or lacked a square-wave capnograph tracing, or if there was airway obstruction (e.g. oxygen desaturation < 90%, abnormal thoraco-abdominal movements, or obstructive noises or no rise of chest at all), inadequate ventilation (an inability to deliver a minimum of 7 ml.kg-1 tidal volumes, or an audible leak)
Oxygen Desaturation less than 90% | 18 months
  It is a Yes or No outcome measure and it will be measured using the oxygen saturation monitor placed on finger and the reading will be detected on the capnography
Gastric Insufflation | 18 months
  It is a Yes or No outcome measure and auscultation with a stethoscope will be performed over the epigastrium during leak pressure testing to detect the occurrence of gastric insufflation
Manipulation of the Device | 18 months
  the number and type of airway manipulations (gentle advancement, withdrawal of device without removal, jaw thrust, or neck extension) required to maintain airway patency during the case will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman M Alzahem, MD, Principal Investigator — King Saud University

IPD SHARING:
Plan to Share IPD: Undecided